CLINICAL TRIAL: NCT06917196
Title: PROOF OF CONCEPT STUDY ON THE EFFICACY OF INHALATORY TARGETED IMATINIB NANOFORMULATIONS IN PULMONARY HYPERTENSION AND POST-INFLAMMATORY FIBROSIS.
Acronym: PROMPTLY
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Stefano Ghio, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: PROMPTLY
Record Dates: First submitted 2025-03-21; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension (PAH); Lung Fibrosis Interstitial
Keywords: PAH; LFD; Pulmonary arterial hypertension; lung fibrosis desease; XHALIP; imatinib
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The PROMPTLY study is a proof-of-concept research project evaluating the efficacy of XHALIP, an innovative inhalable formulation of Imatinib, in treating pulmonary arterial hypertension (PAH) and post-inflammatory fibrosing lung diseases (LFD).

Main Objective To demonstrate the ability of XHALIP to improve the prognosis of PAH and LFD by reducing pulmonary fibrosis and vascular remodeling.

Key Research Questions Is XHALIP effectively absorbed by pathological lung cells? Does it have a beneficial biological effect on cell proliferation and extracellular matrix deposition? Study Plan Preclinical phase: In vitro tests on cells obtained from patients with PAH and LFD.

Absorption and distribution analysis: In vitro lung tissue models to assess drug penetration and effectiveness.

Biological activity assessment: Evaluating XHALIP's ability to inhibit epithelial-mesenchymal transition and cell proliferation.

Participants Patients aged ≥ 18 years diagnosed with PAH or LFD, either candidates for or recipients of lung transplantation.

Biological samples (bronchoalveolar lavage and explanted lung tissues). Methodology Confocal microscopy and flow cytometry to analyze absorption. RT-PCR and Western Blot to assess biological efficacy. Alveolo-capillary models to test drug release and distribution. The study aims to translate preclinical findings into a potential future clinical trial for the development of XHALIP as a novel inhalation-based therapeutic strategy for rare lung diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years diagnosed with fibrosing lung disease, obliterative bronchiolitis, or PAH, who are candidates for or have undergone lung transplantation.
* Obtaining informed consent for all patients enrolled prospectively and all those enrolled retrospectively at their first clinical occurrence at our center.

Exclusion Criteria:

* Suspected or confirmed diagnosis of pulmonary neoplastic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects are enrolled at the Fondazione IRCCS Policlinico San Matteo hospital in Pavia, at the SC of Pulmonology of the Foundation.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-12-04 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Complete synthesis and characterization of XHALIP for in vitro studies. | two years from the enrollment
  Preparation and stabilization of the dry powder formulation of XHALIP.
Complete synthesis and characterization of XHALIP for in vitro studies. | two years from the enrollment
  Evaluation of XHALIP uptake by various cell types obtained ex vivo from patients with LFD and PAH, as well as transplant recipients (endothelial, epithelial, MC, PASMC, inflammatory effector cells), cultured in vitro and in co-culture systems.
Complete synthesis and characterization of XHALIP for in vitro studies. | two years from the enrollment
  Evaluation of CD44 expression by various cell types obtained ex vivo from patients with LFD and PAH, as well as transplant recipients (endothelial, epithelial, MC, PASMC, inflammatory effector cells), cultured in vitro and in co-culture systems.

SECONDARY OUTCOMES:
Exploration of XHALIP Distribution | two years from the enrollment
  The distribution of XHALIP will be studied in thin lung tissue cultures (Precision Cut Lung Slices Cells, PCLSC) obtained from lung explants of patients with LFD and PAH.
Exploration of XHALIP Distribution | two years from the enrollment
  XHALIP distribution will be explored in a model that replicates the alveolo-capillary microenvironment to analyze its interaction with specific pathological human cells and mucosal/surfactant layers, as well as its ability to cross the alveolo-capillary interface.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy